CLINICAL TRIAL: NCT05810012
Title: Comparison of Analgesic Efficacy of Ultrasound Guided Pericapsular Nerve Group Block Versus Fascia Iliaca Compartment Block in Patients of Hip Fracture
Brief Title: Comparison of Analgesic Efficacy of PENB Block with FICB in Post Operative Hip Fracture Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pain Medicine Department (Other)
Responsible Party: Principal Investigator, Moazzam Ali, Consultant Pain Specialist, Pain Medicine Department
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Comparison PENG versus FICB
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2023-03

CONDITIONS: Post-operative Pain Management; Hip Fracture Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PENG Block Group (Experimental)
  Interventions: Drug: PENG block
- FICB Group (Experimental)
  Interventions: Drug: FICB Block

INTERVENTIONS:
Drug: PENG block — 10ml of 0.125% isobaric bupivacaine injected
  Arms: PENG Block Group
Drug: FICB Block — 20ml of 0.125% isobaric bupivacaine injected
  Arms: FICB Group

SUMMARY:
This study was done to evaluate two different interventions for postoperative pain control in patients undergoing hip surgeries. Fifty patients, divided in two equal groups, were included in the study. Patients in Group P were given pericapsular nerve group (PENG) block while those in Group F were given fascia iliaca compartment block (FICB). Pain score, using Numeric Rating scale as a measurement tool, was assessed at one, six, eighteen and twenty fours after the procedure as a primary outcome. Total tramadol consumption in milligrams was recorded as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* surgical correction of fracture neck of femur under spinal anaesthesia

Exclusion Criteria:

* allergy to local anaesthetics
* bleeding disorders
* morbid obesity with BMI more than 35
* patients of chronic pain
* drug addiction
* psychiatric issues

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Pain score using Numeric Rating scale | 24 hours
  Pain scored assessed after completion of surgery at one, six, eighteen and twenty fours

SECONDARY OUTCOMES:
Total Tramadol consumption | 24 hours
  Total Tramadol consumption In twenty four hours

CONTACTS AND LOCATIONS:
Overall Officials: Moazzam Ali, Principal Investigator — Pain Medicine Department
Locations (1):
- Pain Medicine Department, Lahore, Pakistan